Effect of Laughter Yoga on Mental Symptoms Frequency and Level of Cortisol

14/01/2019

Fatma Özlem Öztürk\_RN, Ph. D., Ankara University Faculty of Nursing

Department of Nursing Altindag, Ankara-Turkey, fozlemozturk@gmail.com

Ayfer TEZEL RN, Ph.D. Professor Ankara University Faculty of Nursing

Department of Nursing Altindag, Ankara-Turkey

None conflict of interest statement

Please address all correspondence in regard to this article to: F. Özlem Öztürk, Ph. D., Academician, Ankara University, Faculty of Nursing, Department of Nursing, Altindag, Ankara-Turkey.

E-mail: <u>foozturk@ankara.edu.tr</u>

fozlemozturk@gmail.com

Tel: 90-3123191450-1125

## Informed Consent Form (LAUGHTER YOGA GROUP)

Name of the Study: Effect of Laughter Yoga on the Prevalence of Psychic Symptoms and Salivary Cortisol

Easy to understand the name of the study: Laughter yoga applied and not applied to the group's mental status and the levels of cortisol known as stress hormone evaluation Research Place: Ankara University Faculty of Health Sciences

## General Information

One of the new applications in complementary medicine is laughter yoga. Laughter of laughter, in 1995, a medical doctor in India, Dr. Madan Kataria has developed. Laughter yoga is a non-invasive and non-pharmacological treatment method. Laughter of laughter has positive effects on mental health. It is reported that depression provides a reduction in anxiety, is an effective strategy for coping with stress and improves quality of life. It is also stated that laughter has many physiological effects. Our body's laughter; increase in respiratory rate, increase in oxygen saturation in the blood, increase in heart rate, decrease in blood pressure, decrease in muscle tension, decrease in stress hormones such as adrenaline, noradrenaline, cortisol, give rise to physical reactions such as improvement in immune system functions and mental processes.

One session of laughter yoga; hand whipping and warm-up exercises, deep breathing exercises, childish games and laughter exercises. One session of laughter yoga takes about 40 minutes. In this study, 8 sessions of laughter yoga will be applied twice a week for 4 weeks. Objective: The aim of this study was to investigate the effects of laughter yoga on mental health symptoms and cortisol levels.

Under the leadership of the researcher, you will have 8 sessions of laughter yoga in total with two sessions per week for four weeks. Each of you will receive a saliva sample for measurement of cortisol sixteen times during 8 sessions before and after all laughter yoga starts. After the latest laughter yoga session, a questionnaire will be applied again. Laughter yoga sessions will be held in a suitable day and class according to your schedule. You will be given saliva tubes before and after the laughter yoga session. You will be asked to soak the roll cotton material inside the tubes with saliva for at least 1 minute and place them in the tube again. Saliva samples will be taken to the hungry wife at 08.00-08.40 in the morning. Your participation in the research is entirely at your discretion and you have the right to refuse to participate in the research. You can quit research at any time. You will not take any financial responsibility for participating in this research. You will not be charged any further. The information to be taken from you will only be used in the aforementioned study. Your credentials and the information you provide will be kept confidential. Failure to participate in the study will not affect your education process positively or negatively. You can ask F. Özlem ÖZTÜRK when you have a question about the research. Thank you for your participation.

I .. read and understood the information written above. I was informed verbally about the research. I agree to participate in the research. History: ..../...../...........

## (CONTROL GROUP)

Name of the Research: Evaluation of the Effect of Laughter Yoga on the Frequency of Psychiatric Symptoms and Salivary Cortisol Level in 1st Grade Students of Nursing Department

Easy to understand the name of the study: Laughter yoga applied and not applied to the group's mental status and the levels of cortisol known as stress hormone evaluation Research Place: Ankara University Faculty of Health Sciences

## General Information

One of the new applications in complementary medicine is laughter yoga. Laughter of laughter, in 1995, a medical doctor in India, Dr. Madan Kataria has developed. Laughter yoga is a non-invasive and non-pharmacological treatment method. Laughter of laughter has positive effects on mental health. It is reported that depression provides a reduction in anxiety, is an effective strategy for coping with stress and improves quality of life. It is also stated that laughter has many physiological effects. Our body's laughter; increase in respiratory rate, increase in oxygen saturation in the blood, increase in heart rate, decrease in blood pressure, decrease in muscle tension, decrease in stress hormones such as adrenaline, noradrenaline, cortisol, give rise to physical reactions such as improvement in immune system functions and mental processes.

One session of laughter yoga; hand whipping and warm-up exercises, deep breathing exercises, childish games and laughter exercises. One session of laughter yoga takes about 40 minutes. In this study, 8 sessions of laughter yoga will be applied to the experimental group twice a week for 4 weeks. No laughing yoga will be applied to the control group. Objective: The aim of this study was to investigate the effects of laughter yoga on mental health symptoms and cortisol levels.

As a result of our research, you will receive a saliva sample for the measurement of cortisol level six times a week for 8 sessions twice a week on the days and hours of saliva samples taken from the experimental group. Saliva samples will be taken by F. Özlem ÖZTÜRK at Ankara University Faculty of Health Sciences on the same days and hours as the experimental group at 08.00-08.40. You will be asked to soak the roll cotton material inside the tubes with saliva for at least 1 minute and place it back in the tube.

Laughter yoga will not be applied to you. After the research is completed you will be able to apply the laughter yoga.

Your participation in the research is entirely at your discretion and you have the right to refuse to participate in the research. You can quit research at any time. You will not take any financial responsibility for participating in this research. You will not be charged any further. The information to be taken from you will only be used in the aforementioned study. Your credentials and the information you provide will be kept confidential. Failure to participate in the study will not affect your education process positively or negatively. You can ask F. Özlem ÖZTÜRK when you have a question about the research.

Thank you for your participation.